CLINICAL TRIAL: NCT02910687
Title: Frailty as an INstrument for Evaluation of Elderly Patients With Non ST ElevationMyocardial Infarction (NSTEMI) - 5 Year Follow up (FINE75+5)
Brief Title: FINE75+: 5 Year Follow up
Acronym: FINE75+5
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Niklas Ekerstad, MD, PhD, Linkoeping University
Other Study IDs: FINE75+5
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-03

CONDITIONS: Non ST Elevation Myocardial Infarction (NSTEMI); Frailty
Keywords: Non ST Elevation Myocardial Infarction (NSTEMI); Elderly; Frailty; Prognostic value
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NSTEMI75+: Patients, 75 years old or older, with Non ST Elevation Myocardial Infarction (NSTEMI)
  Interventions: Other: This is an observational study

INTERVENTIONS:
Other: This is an observational study

SUMMARY:
In the FINE 75+ study, 307 Non ST Elevation Myocardial Infarction (NSTEMI) patients, 75 years old or older, were included between September 2009 and June 2010. The purpose of this observational study (FINE75+5) is to describe these patients, especially regarding the following variables: cardiovascular risk, co-morbidity and frailty, and to assess the prognostic value of frailty on 5-year outcomes. We hypothesize that frailty is independently associated with 5-year mortality.

DETAILED DESCRIPTION:
The term frailty denotes a multi-dimensional syndrome characterized by increased vulnerability and decreased physiologic reserves. Frailty stratification predicts a patient's risk of death and need for institutional care. The construct is well validated, but there is not one single accepted operational definition. The CSHA Clinical Frailty Scale (CFS) is a 7-point scale relying on clinical judgement. It is a global clinical measure of biological age, and it mixes co-morbidity, disability and cognitive impairment.Though frailty instruments so far mainly have been used in a geriatric context, it has been pointed out as relevant for cardiologic patients as well, e.g. regarding risk stratification for elderly patients with NSTEMI.

In the FINE 75+ study, 307 Non ST Elevation Myocardial Infarction (NSTEMI) patients, 75 years old or older, were included between September 2009 and June 2010. We reported importance of frailty for short-term (1 month) and medium-term outcome (1 year) in a NSTEMI population (Ekerstad et al. 2011, Ekerstad et al. 2013). However, there are no published data on the importance of frailty on longer-term outcome. Information on long-term prognosis may substantially improve informed decision making in elderly patients with NSTEMI, with acute potentially harmful treatments aiming at improved long-term prognosis.

The purpose of this study is to describe patients, 75 years old or older, with NSTEMI especially regarding the following variables: cardiovascular risk, co-morbidity and frailty, and to assess the prognostic value of frailty on 5-year outcomes.For the purpose of the current analysis all patients included in the final FINE 75+ study will be followed over 5 years from hospital admission. We hypothesize that frailty is independently associated with 5-year mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients included in the FINE 75+ study population between October 2009 and June 2010. Patients, 75 years old or older, with diagnosed NSTEMI, and cared for at one of the following hospital care units: cardiology, acute medicine, geriatrics, other internal medicine unit.

Exclusion Criteria:

* Not willing to participate. Non-evaluable patient due to communication problems and insufficient clinical information for the judgement of frailty.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients included in the FINE 75+ study population between October 2009 and June 2010. They were consecutive evaluable patients, 75 years old or older, with diagnosed NSTEMI,and cared for at one of the following hospital care units in the University Hospital ofLinköping and the County Hospitals in Trollhättan (NÄL-Uddevalla) and Jönköping (Ryhov): cardiology, acute medicine, geriatrics, other internal medicine unit.
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
All-cause mortality at 5 year follow up | 5 years

SECONDARY OUTCOMES:
Rehospitalisation for myocardial infarction, stroke, other cardiovascular disease, bleeding complication, fracture, cancer or other diagnosis. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Ekerstad, MD, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linkoeping University Hospital, Linköping, Ostergoetland, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ekerstad N, Swahn E, Janzon M, Alfredsson J, Lofmark R, Lindenberger M, Carlsson P. Frailty is independently associated with short-term outcomes for elderly patients with non-ST-segment elevation myocardial infarction. Circulation. 2011 Nov 29;124(22):2397-404. doi: 10.1161/CIRCULATIONAHA.111.025452. Epub 2011 Nov 7. PMID 22064593
- [Background] Ekerstad N, Swahn E, Janzon M, Alfredsson J, Lofmark R, Lindenberger M, Andersson D, Carlsson P. Frailty is independently associated with 1-year mortality for elderly patients with non-ST-segment elevation myocardial infarction. Eur J Prev Cardiol. 2014 Oct;21(10):1216-24. doi: 10.1177/2047487313490257. Epub 2013 May 3. PMID 23644488